CLINICAL TRIAL: NCT04295174
Title: KIDSTAGE- Staging of Kidney Cancer Using Dual Time PET/CT and Other Biomarkers
Status: Completed | Type: Observational
Sponsor: Odense University Hospital (Other)
Responsible Party: Principal Investigator, Louise Geertsen, Medical doctor, Odense University Hospital
Other Study IDs: S-20160005
Record Dates: First submitted 2020-03-03; First posted 2020-03-04 (Actual); Last update posted 2020-03-04 (Actual); Status verified 2020-03

CONDITIONS: Carcinoma, Renal Cell
Keywords: circulating tumor DNA
MeSH Terms: conditions — Carcinoma, Renal Cell

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Collection of tumorsamples and blodsamles before and after nephrectomy in patients with renal cell carcinoma
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
Kidney cancer is a highly malignant disease with 950 new cases every year in Denmark. Diagnosis and treatment of kidney cancer patients presents many challenges because that early stages of the disease are often asymptomatic and the disease is thus often at advanced stage or even metastatic when discovered. Metastasis is a predictor of bad prognosis, because the presence of metastases excludes the possibility of curative treatment (surgery). Systemic (medical) treatment is used for metastatic disease. It is of increasing importance to monitor how patients are responding to the treatment and switch to a different product if the tumor is not responding. Improved methods for detection of metastatic lesions would be of great advantaged for the clinicians in order to select the optimal treatment strategy for the patients.

In the present study we aim to identify tumor markers in the blood and more specific we want to investigate whether circulating tumor-DNA can be used as a biomarker for monitoring the development of the disease during and after treatment. We want a better understanding of the tumor's heterogeneity and development. Furthermore we want to evaluate the diagnostic value of dual time FDG- PET/CT for the detection of bone and lymph node metastases in patients with kidney cancer

DETAILED DESCRIPTION:
Background Renal cell carcinoma (RCC) represents 2-3% of all malignancies, and the European prevalence is approximately 84,400 cases per year [1]. In Denmark 950 new cases of Kidney Cancer (KC) are diagnosed per year, and the incidence is increasing annually. KC is more common in men than in women and the cancer debuts most frequently in the age of 60-70 years [2]. Early stages of KC are often asymptomatic and the disease is thus often at advanced stage or even metastatic when discovered. Metastases including lymph node metastases are a predictor of bad prognosis. Surgical removal of cancerous lymph nodes has been shown to improve response to systemic treatment and prolong survival [3], but the current methods for detection of especially lymph node metastases are insufficient. Improved methods for detection of metastatic lesions at the time of diagnosis would be of great help for the clinicians who have to select the optimal treatment strategy for the patients. Surgery is the only curative treatment and also the predominant choice of treatment when possible. Systemic treatment is only used in case of metastatic disease. Metastatic KC is generally non-responsive to chemotherapeutics and radiation therapy [2], but a range of other systemic treatment options has been developed over the last decade. This means that it is of increasing importance to monitor how patients are responding to the selected treatment and switch to a different product if the tumor is not responding. The number of patients with KC identified by chance has increased along with an increasing use of routine imaging for a number of others disorders [4]. It is still likely that new and improved methods for early detection of cancer would improve the survival in KC patients.

PET/CT:

Positron Emission Tomography (PET) combined with computed tomography (CT) is a well-established method of diagnosing and staging several types of cancer. 2-deoxy-2-[18F]fluoro-D-glucose (FDG) is the most common PET tracer used in oncologic studies. PET/CT is not a standard modality in the diagnosis and staging of RCC [5]. The sensitivity as to detection of the primary tumor is hampered by the physiological excretion of FDG in the urine. Furthermore, histological characteristics of the tumor such as grade and expression of glucose transporters can affect the FDG uptake negatively [6]. However, PET/CT performs well in detection of extra-renal metastases [7, 8] and proved to be of prognostic value in recurrent RCC [9].

FDG is accumulated in cells with increased glycolysis, in particular cancer cells. FDG accumulation is not specific to tumors and is also seen in benign processes such as inflammation and infection. This makes it diﬃcult to distinguish malignant neoplastic lesions from the benign ones [10]. In recent years the concept of dual-time point (DTP) imaging has evolved. The increase in FDG uptake seems to continue for hours after injection in malignant tissue whereas FDG uptake in normal or inflamed tissue reaches maximum uptake earlier and declines thereafter. Thus, late imaging is thought to result in increased FDG uptake, decreased blood and urine activity and, thus, a better target-to-background ratio and, therefore, a higher sensitivity [11]. Several studies using DTP PET/CT have been performed on tumors in the breast, liver, lung, and prostate. Results indicate that the pattern and rate of FDG uptake over time vary considerably between malignant and benign processes and that DTP PET/CT allows for distinction between them [12,13]. Hitherto, the use of DTP imaging in RCC was scantily reported. A recent paper considered the value of DTP imaging of the primary renal tumor but not of the metastases [14].

Circulating tumor DNA There is a general and increasing interest in circulating cancer biomarkers because they might constitute representative readouts of both primary tumor and metastatic deposits. Furthermore, circulating markers may provide a tool for monitoring response to systematic adjuvant therapies even after the primary tumor has been removed. Promising results have been obtained for blood-born cell free DNA (cfDNA) which can be isolated from a simple blood sample, often referred to as a liquid biopsy. In contrast to tissue biopsies, detection of cfDNA from peripheral blood is a minimally invasive way to monitor the disease during treatment and follow-up.

cfDNA is assumed to be released from most or all of the cells in the body and is present in healthy as well as sick individuals. Several studies report that specific alterations from tumor tissue is mirrored in cfDNA and that it is thus possible to discriminate circulating tumor DNA (ctDNA) from normal cfDNA. Studies applying sequencing of somatic mutations in well-known cancer driver genes like TP53, PIK3CA, and KRAS have been reported and promising results have been obtained for using these markers for early detection of recurrence in colorectal cancer [15] breast cancer [16] and lung cancer [17]. A drawback in this approach is that a considerable fraction of solid tumors do not contain mutations in these candidate genes. This challenge can be met by using next generation sequencing of tumor tissue to identify tumor-specific alterations which may then be monitored in plasma. Two recent studies applied low-coverage whole genome sequencing of tumor tissue to detect tumor-specific breakpoint and subsequently used PCR-based assays targeting these breakpoints to detect and monitor ctDNA burden in patients with colorectal cancer [18] and breast cancer [19]. The method proved to be highly sensitive and specific in the discrimination between patients with and without recurrence, and they were able to detect metastatic recurrence with a lead time of 10 and 11 months, respectively, compared to conventional methods. Furthermore, Reinert and co-workers [18] also demonstrated that the level of ctDNA varied with administration of therapy and that ctDNA may be used as a tool to monitor treatment response. One of the most significant and early hallmarks of tumors are genomic instability which represents a driving force behind the development of therapy resistance and metastasization. Genomic instability is one of the major challenges in the systemic treatment of cancer because the resulting tumor heterogeneity is not only difficult to uncover, but also dynamic and thus challenging to monitor in time. Genetic profiles of tumors are commonly obtained from tissues biopsies, however these may not reveal relevant tumor heterogeneity and the invasiveness of the procedure makes them unsuitable for sequential monitoring during disease progression. ctDNA may represent a minimally invasive way to monitor not only tumor load but also tumor heterogeneity and evolution towards metastasis.

Hypotheses

1. Increase in FDG uptake continues for hours after injection. Late imaging (DTP FDG PET/CT) should result in increased FDG uptake, decreased blood and urine activity and, thus, a better lesion-to-background ratio. By combining this with the pathological report it might be possible to get a better staging of the kidney cancer patients.
2. Tumor burden, heterogeneity and dissemination is reflected in circulating tumor-DNA (ctDNA), which can be measured in a simple blood sample. Analysis of ctDNA can be expected to provide information about changes in tumor load before - and during treatment, and in patients with metastatic disease and during their treatment.

Aim The primary purposes of these prospective trials are to investigate the use of DTP FDG PET/CT in staging of lung, bone- and lymph node metastasis in patients with KC and to investigate if ctDNA can be used as a tool for assessment of tumor load, tumor heterogeneity, dissemination, for monitoring during treatment and disease progression in KC patients.

KIDSTAGE I: DTP FDG PET/CT for detection of lung-, bone- and lymph node metastases in patients with KC Population All patients diagnosed with KC in The Urological Department and in The Oncological Department of OUH are eligible for enrolment in the study.

Inclusion criteria:

* KC patients at Urological- and Oncological departments of OUH
* Written consent
* Able to speak and understand Danish

Exclusion criteria:

* Patients below 18 years of age
* Patients with mental impairment
* Withdrawal of consent
* Other malignancy Methods Patients included in the study will have a DTP FDG-PET/CT scan. The scans will be performed before the nephrectomy/administration of oncological treatment. The Department of Nuclear Medicine perform the scans with acquisition 1 and 3 hours after administration of the FDG tracer. Images are interpreted by a specialist in nuclear medicine. Images are interpreted based on visual evaluation with supplementary measurements of Standardized uptake values (SUV). SUVmax will be determined for both the early and late acquisition (SUVearly and SUVlate). A retention index (RI) will be calculated as (SUVlate - SUVearly)/SUVearly.

Primary target imaging variables will be "metastases to the lungs" (yes/no), "metastases to lymph nodes" (yes/no) and "metastases to bone" (yes/no). Secondary analyses will be lesion-based. In according to lymph node detection, lesion-based describe each lymph node group. Activity in regional lymph nodes will be recorded according to their location; "renal hilus (dx/sin)", "retroperitoneal para aortic" and "para cavale"[2]. During the nephrectomy the lymph nodes from the above mentioned stations will be removed and placed in separate containers marked as: "renal hilus dx.", "renal hilus sin.", "para aortic" and "para cavale". Pathologists will examine the tissue samples. The results of the PET/CT will not be available to the pathologist. The results of the PET/CT will be compared to results of histological examination (Gold Standard) and sensitivity, specificity, positive and negative predictive value will be calculated.

Results regarding lung and bone metastases will be compared to the results of the diagnostic CT scan of thorax/abdomen that is already made for each patient as a part of the standard examination program. In case of agreement between the scans, the patient will proceed to clinical treatment as usual. In case of disagreement between the modalities concerning bone, a Magnetic Resonance Imaging (MRI) will be performed of the lesion of interest. If the results after MRI are still inconclusive a bone biopsy with emphasis on getting marrow tissue as well as bone matrix, will be performed. This will in many cases not be possible due to the size of the lesion and in these cases MRI will serve as reference standard.

All results will be coded and given an ID according to patient´s CPR number using the RedCap informatic coding system.

KIDSTAGE II: Circulating biomarkers in KC and tumor heterogeneity Population All patients with KC at The Urological Department of OUH who undergo surgery and all patients admitted at the departments at OUH who undergo kidney biopsy for suspect renal tumor will be considered potentially suitable for the enrolment.

Inclusion criteria:

* Patients with KC without metastases treated at Urological Department of OUH
* Written consent
* Able to speak and understand Danish Exclusion criteria
* As in KIDSTAGE I Methods Sample collection A blood sample (20 ml) will be taken pre-operatively from each patient participating in the study. The sample collection will be repeated at the first postoperative day while the patient is still hospitalized and after 2 weeks, 3, 6 and 12 months. All samples will be coded and given an ID according to patient´s CPR number using the RedCap informatic coding system. Furthermore, a biopsy of the tumor on the surgically removed kidney will be sent to the Department of Pathology. The tumor sample will also be coded according to RedCap. Sizes of the histological specimen as ported for the study will be of 5 mm x 5 mm x 5mm.

Sample analysis The blood samples will be delivered to the Department of Clinical Genetics at OUH and will be centrifuged to separate plasma from blood cells and both fractions will be stored at -80C. Isolation of DNA from tumor tissue, lymphocytes and plasma (cfDNA) will be performed using commercial kits.

KIDSTAGE IIa: DNA isolated from tumor tissue will be subjected to low coverage (approximately 1-3 X) whole genome sequencing with 2 X 100 paired end reads and long inserts. Sequencing will be performed using an Illumina HiSeq1500 located at Department of Clinical Genetics in Odense. The large somatic mutations will be filtered to avoid known germline copy number variations and will finally be validated as somatic mutations by personalized assay of DNA from lymphocytes. A considerable number of large somatic mutations are expected to be identified in all tumors using this pipeline. A smaller number of 2-3 mutations from each tumor will be implemented in a personalized PCR set-up covering the breakpoints of identified somatic mutations. Quantification will be performed using digital PCR and a number of housekeeping genes will be used for normalization. The assays will be applied to 1) plasma samples to detect and quantify ctDNA and 2) DNA isolated from the cell fraction of the blood sample in order to validate that the mutations are somatic.

KIDSTAGE IIb: For 20 patients tumor heterogeneity will be studied by isolating DNA from 4 independent biopsies from the resected primary tumor and from normal tissue (normal blood cells). Whole exome sequencing is performed at 100X coverage, suspected somatic point mutations are called by comparing sequences from tumor and normal tissue [20] validation and accurate estimates of allele frequencies are obtained by ultra deep (>1000X) targeted sequencing of suspected mutations. The subclonal structure is deciphered by bioinformatics analysis. This procedure was successfully applied in one of our previous studies [21]. In order to determine to what extent the heterogeneity is reflected in ctDNA, the ultra deep sequencing will also be performed on the ctDNA from the same patient.

Sample storage discharge Purified samples will be anonymously stored in a research biobank for a maximum period of 10 years from collection. After that time, all samples will be destroyed. In case of performance of further analyses on the samples, than to those illustrated in the present protocol, both for the aims of the present study or for new studies, explicit allowance will be previously requested to the ethical committee and to the respective organs in charge for these purposes

KIDSTAGE III: Circulating biomarkers in metastatic KC and tumor evolution Population All patients with metastatic KC treated at The Oncological Department of OUH will be considered potentially suitable for the enrolment.

Inclusion criteria:

* Patients with histologically verified and metastatic KC treated in Oncological Department of OUH
* Written consent
* Able to speak and understand Danish Exclusion criteria
* As in KIDSTAGE I Methods Sample collection For patients with metastatic KC in the "good" and "intermediate" prognosis groups the first line treatment is Pazopanib 800 mg given daily. This is given continuously until progression. Evaluation of treatment response is performed by a clinical control at the Department of Oncology every 4 week and with a CT-scan every 3 month. For patients in the poor prognosis group and for patients with not clear-cell-type the first line treatment is Sunitinib 50 mg. This is given daily for 4 weeks and then a break for 2 weeks. Evaluation of treatment response is performed by a clinical control at the Department of Oncology every 6 week and with a CT-scan every 3 month.

A blood sample (20 ml) will be taken from each patient before initiating the oncological treatment. Sample collection will be repeated after 2 weeks, 3, 6 and 12 months. All samples will be coded and given an ID according to patient´s CPR number using the RedCap informatic coding system. An ultrasound guided biopsy of the primary tumor and the metastases will be taken and sent to the Department of Pathology, OUH. This is a standard procedure for patients with metastatic disease, who are planned for oncological treatment. The tumor sample will also be coded according to RedCap.

Sample analysis KIDSTAGE IIIa: As in KIDSTAGE IIa KIDSTAGE IIIb: For 20 patients tumor evolution is studied by isolating DNA from biopsies from primary tumor, metastasis and normal cells. Like in IIb whole exome sequencing, variant calling and ultra deep sequencing are performed. The genomic evolution from primary tumor tp metastasis is deciphered by bioinformatics analysis, as we reported previously [22,23]. In order to determine to what extent this evolution is reflected in ctDNA, ultra deep sequencing will be performed on ctDNA too.

Sample storage discharge As in KIDSTAGE II Sample size Annually 100-120 patients diagnosed with KC undergo surgery at The Urological Department of OUH and 70-80 patients with metastatic KC are treated at The Oncological Department of OUH. Approximately 75 patients will be a realistic no of patients to enroll in the overall study. Since this is an explorative study and no other larger studies have investigated this, it has not been possible to make power calculations for the sample size.

Feasibility The patients will be enrolled in the study when a diagnosis of KC has been made in The Urological Department or in The Oncological Department of OUH. Contact to the patients will be facilitated by Louise Geertsen. Collection of blood samples will be performed by technicians or by Louise Geertsen.

Sequencing, data analysis and ddPCR will be performed at the Department of Clinical Genetics at OUH. The department has the Illumina HiSeq technology and computing power for Next Generation Sequencing (NGS) and has implemented NIPT as a clinical analysis. Prof. Torben A. Kruse and his team has years of experience with NGS and cancer research, and comprehensive technical and bioinformatical knowledge including detection of breakpoints and copy number variations from NGS has been obtained[20,21,22,23]. The DTP PET/CT scans will be performed at The Department of Nuclear Medicine, OUH. The department has years of experience in performing and interpreting FDG PET/CT and DTP FDG PET/CT [24,25,26]. The images will be interpreted by Jane Simonsen, PhD and consultant at The Department of Nuclear Medicine or a substitute for her. Histological examination of tumor biopsies will be facilitated by our collaboration partner Niels Marcussen, professor and consultant at the Department of Pathology.

Ethics

Ethical aspects to be considered in KIDSTAGE I:

Most patients will be 60 years of age or older at the time of diagnosis, and few if any will be younger than 50 years. In Denmark the theoretical lifetime risk of dying due to cancer is approximately 25% for a 25-year old subject. For each Sv the risk of inducing cancer is increased by 5% compared to the overall risk in the population. By exposure of a radiation dose of 28 mSv = 0.028 (0.03) the risk increases by 5% * 0.03 = 0.2% after participation in the study. However, the risk is age-dependent and due to the national guidelines [27] the present project can be considered as a category IIb research project, because all patients will be above the age of 50 years. For a research project of this category to be approved, the benefits of the project should be expected to be "directed towards diagnosis, cure or prevention of disease" - which is exactly the case for the present study. The increased risk due to radiation has to be held up against the potential benefit for the patient participating in the study and for future patients. The potential benefit for the patient participating in the study is foremost a possibly better staging of the disease. Furthermore, if the study on lymph nodes shows trends towards usefulness in detecting lymph node metastases, then this could be of immense benefit for future patients.

Ethical considerations that apply in KIDSTAGE II and III: When we determine the DNA sequence of the entire genetic material, there is a small risk of finding genetic defects in the genome. Some genetic defects can cause hereditary diseases and can affect the health of the patient and the patient´s family. In some cases, it is possible to treat or even prevent the disease caused by that gene defect and in other cases it is not. In the written information that the patient is given, this risk will be mentioned and the patient is given the opportunity to decide how much information they want to know of their own genetic material. In situations where we find a defect in the genome that can cause disease in the long term, and where the patient wanted to be informed, the patient will be invited for an interview in the clinic. During this interview, there will be a genetic counsellor present. The genetic counsellor will inform the patient about what the information means for the patient and the patient's family.

The above mentioned studies (Project-ID S-20160005), the patient information sheets and the informed consent form was approved by The Regional Scientific Ethical Committees for Southern Denmark February 4, 2016 and by the local data protection agency "Datatilsynet" in October 2016 with the Professor MD Lars Lund as main supervisor for PhD student Louise Geertsen. The trial will be conducted in accordance with Good Clinical Practice, Declaration of Helsinki.

ELIGIBILITY:
Inclusion Criteria:

* KC patients at Urological- and Oncological departments of OUH
* Written consent
* Able to speak and understand Danish

Exclusion Criteria:

* Patients below 18 years of age
* Patients with mental impairment
* Withdrawal of consent
* Other malignancy

Min Age: 18 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: patients diagnosed with renal cell carcinoma in The Urological Department and in The Oncological Department of OUH are eligible for enrolment in the study
Sampling Method: Non-Probability Sample
Enrollment: 70 (Actual)
Dates: Start 2018-01-01 (Actual); Primary Completion 2020-01-01 (Actual); Study Completion 2020-01-01 (Actual)

PRIMARY OUTCOMES:
circulating tumor DNA in patients with renal cell carcinoma | 3 years
  investigating if circulating tumor DNA can be used to monitor tumor burden and disease progression in patients with renal cell carcinoma
Dual time point FDG PET/CT in patients with renal cell carcinoma | 1 year
  investigating if Dual time point FDG PET/CT can be used in staging of renal cell carcinoma

CONTACTS AND LOCATIONS:
Overall Officials: Lars Lund, MD, DMSci, Principal Investigator — Professor, Consultant Urology, Department of Urology, Odense University Hospital
Locations (1):
- Odense University Hospital, Odense C, Odense, Denmark